CLINICAL TRIAL: NCT01379924
Title: Young Parents Program, Project Connect
Acronym: YPPProCon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joanne Cox, Associate Chief, Division of General Pediatrics; Medical Director, Boston Children's Primary Care, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5 APHPA002033-10-00
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Adolescents; 18 and Under When Child Was Born for Mothers; 25 and Under When Child Was Born for Fathers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young Parents Program plus Parenting/Life Skills modules (Experimental): In addition to receiving standard medical and social services for young parents and their children, patient takes part in 5 one on one modules during the first year of child's life aimed at educational attainment, budgeting, child development, safety in the home and substance abuse.
  Interventions: Behavioral: Parenting/Life Skills Intervention
- Young Parents Program usual care (Active Comparator): Patients receive regular standard of care without modules.
  Interventions: Other: Teen-tot medical home

INTERVENTIONS:
Behavioral: Parenting/Life Skills Intervention — Modules adapted from the Ansell-Casey Life Skills Assessment Curriculum, the Women's Negotiation Project Curriculum for Teen Mothers and the Nurturing Curriculum. Goal is to help teen mothers develop positive parenting skills, decrease repeat pregnancy and acquire skills of daily living. The series of five, one-hour long, structured, one-on-one interactive modules aims to help teens build positive, empathetic relationships with their children, while enhancing self-efficacy and increasing the sense of self- worth for parents and children. Domains addressed include child development/discipline, safety, house/money management, social relationships, career planning, substance abuse and community and interpersonal violence.
  Arms: Young Parents Program plus Parenting/Life Skills modules
Other: Teen-tot medical home — Medical, mental health, and social services provided to teen parents and their children
  Arms: Young Parents Program usual care

SUMMARY:
1. Specific Aims

1. To evaluate the effects of life skills/parenting groups that are embedded within a comprehensive multidisciplinary clinic for adolescent parents (the Young Parents Program), using a randomized control design. Specifically, the effect of group participation on the following adolescent parent outcomes will be investigated:

   * Parenting attitudes and skills including empathy, non-violent discipline, role appropriateness and developmentally appropriate expectations.
   * Skills of daily living, social relationships, and work/study at follow-up, as measured by the Ansell-Casey Life Skills Assessment Scale.
   * Depression and perceived social support using the CESD-C and Duke Social Support scale.
   * Repeat pregnancy rates at 12 and 24 months after first delivery.
2. To evaluate the overall Young Parents Program service delivery as required by the Office of Adolescent Pregnancy Programs (project funder) using a cross cutting evaluation of health services utilization, social needs and work/educational outcomes.

DETAILED DESCRIPTION:
The Young Parents Program (YPP), a specialty clinic within Children's Hospital Primary Care Center, provides comprehensive medical care, mental health services, and advocacy to high risk, urban teen parents and their young children through a teen-tot model. YPP serves 152 teenage mothers and their babies annually with a multi-disciplinary team knowledgeable in the medical, social, and developmental issues of adolescence and early childhood. Project Connect is an evaluation of both the medical and social services provided by YPP and a randomized controlled trial of an intensive educational arm of YPP.

YPP serves the population that economically, ethnically, and geographically represents the highest rates of subsequent pregnancies and the greatest risk for poor birth outcomes. The staff of physicians, nurse practitioners, social workers, and nurse consists of experienced professionals work with parents, adolescents, and children. YPP has cooperative relationships with Boston area education and job training sites, Early Intervention Programs, the Massachusetts Department of Revenue, community agencies, mental health services, and teen living programs.

By providing an integrated family based comprehensive medical home and a randomized controlled trial of intensive parenting/life skills training, Project Connect enhances teen parents' connections to child, family, peers, partners, medical care, and mental health. Medical care, home visiting, child/adolescent health services, mental health, and fathers' programming are all linked into a continuous program. Goals of the intensive intervention are to enhance parenting and life skills, help participants optimize family interactions, and build self-efficacy.

Project Connect brings together YPP at Boston Children's Hospital (BCH), Healthy Baby/Healthy Child (HB/HC) nurse home visiting program and Families First, a parenting education agency, to provide a state-of-the art model of care for parenting teens in Boston. The model builds on lessons learned and strengths of each program, adding critical new elements of randomized control trial of parenting/life skills modules, and home visiting. Prenatal services will encourage breast-feeding, and support infant care and parenting. YPP provides a medical home with coordinated, continuous health care services, psychosocial support, parenting/life skills modules and individual services for teen mothers and fathers. Integrated fathers' services emphasize male parenting roles, communication, life skills training, violence prevention and positive youth development.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to speak and read in English
* Mothers must be 18 or under when baby is born
* Fathers must be 25 or under when baby is born
* Child must be seen in YPP
* Willing to complete computer surveys 6 times over 36 months
* Ability to complete computer assisted data collection

Exclusion Criteria:

* If parent does not have custody of children
* If children are no longer receiving care at YPP

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Cox, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hosptial, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cox JE, Harris SK, Conroy K, Engelhart T, Vyavaharkar A, Federico A, Woods ER. A Parenting and Life Skills Intervention for Teen Mothers: A Randomized Controlled Trial. Pediatrics. 2019 Mar;143(3):e20182303. doi: 10.1542/peds.2018-2303. Epub 2019 Feb 12. PMID 30755464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a teen-tot program (Young Parents Program) within a pediatric hospital. Eligibility criteria included maternal age <19 years at delivery and infant age <12 months old. At the first infant visit, every patient seen was asked to enroll in the study by trained program staff. assignment.
Pre-assignment Details: Of 152 eligible patients who received care in the Young Parents Program who were invited to participate in the randomized trial, 12 declined to participate and were never enrolled into the study, but continued to receive care in the program.
Groups:
- Young Parents Program Plus Parenting/Life Skills Modules: These modules were developed using the Ansell-Casey Life Skills Assessment Curriculum and The Women's Negotiation Project Curriculum for Teen Mothers. The Nurturing Curriculum has been shown in our past program to be associated with increased parenting skills, maternal self-esteem and decreased life hassles. The nationally recognized Nurturing Curriculum is integrated with the Ansell-Casey life skills Curriculum and The Women's Negotiation Project Curriculum to help teen mothers develop the skills and communication needs of daily living. The series of five, one-hour long, structured, one-on-one interactive modules aims to help teens build positive, empathetic relationships with their children, while enhancing self-efficacy and increasing the sense of self- worth for parents and children. Domains addressed include child development/discipline, safety, house/money management, social relationships, career planning, substance abuse and community and interpersonal violence.
- Young Parents Program Usual Care: Patients receive regular standard of care without modules.
  No intervention
Period: Baseline
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Started | 72 | 68
Completed | 72 | 68
Not Completed | 0 | 0
Period: 12-month Assessment
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Started | 72 | 68
Completed | 62 | 55
Not Completed | 10 | 13
Period: 24-month Assessment
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Started | 62 | 55
Completed | 55 | 52
Not Completed | 7 | 3
Period: 36-month Assessment
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Started | 55 | 52
Completed | 52 | 48
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Young Parents Program Plus Parenting/Life Skills Modules: Patient takes part in modules that were developed using the Ansell-Casey Life Skills Assessment Curriculum and The Women's Negotiation Project Curriculum for Teen Mothers. The Nurturing Curriculum has been shown in our past program to be associated with increased parenting skills, maternal self-esteem and decreased life hassles. This curriculum is integrated with the Ansell-Casey life skills Curriculum and The Women's Negotiation Project Curriculum to help teen mothers develop the skills and communication needs of daily living. The series of five, one-hour long, structured, one-on-one interactive modules aims to help teens build positive, empathetic relationships with their children, while enhancing self-efficacy and increasing the sense of self- worth for parents and children. Domains addressed include child development/discipline, safety, house/money management, social relationships, career planning, substance abuse and community and interpersonal violence.
- Young Parents Program Usual Care: Those in the control group receive the YPP standard of care including comprehensive multi-disciplinary team medical and mental health support and toddler educational family forums during year 2. No intervention.
- Total: Total of all reporting groups
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care | Total
Number analyzed (Participants) | 72 | 68 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.4 (1.0) | 17.3 (1.2) | 17.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 68 | 140
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latina | 39 | 44 | 83
  Black non-Hispanic | 28 | 18 | 46
  Other non-Hispanic | 3 | 6 | 9
  Not reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rapid Repeat Pregnancy
Description: Number and percent with any repeat pregnancy by each follow-up time point.
Time Frame: 12 months follow-up
Population: Participants with pregnancy data available at 12 months follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Young Parents Program Plus Parenting/Life Skills Modules: Intervention Modules were developed using the Ansell-Casey Life Skills Assessment Curriculum and The Women's Negotiation Project Curriculum for Teen Mothers and the Nurturing Curriculum. The series of five, one-hour long, structured, one-on-one interactive modules aims to help teens build positive, empathetic relationships with their children, while enhancing self-efficacy and increasing the sense of self- worth for parents and children. Domains addressed include child development/discipline, safety, house/money management, social relationships, career planning, substance abuse and community and interpersonal violence. Family planning is discussed at each session.
- Young Parents Program Usual Care: Patients receive regular standard of care without parenting/life skills intervention.
  No intervention
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 62 | 55
Participants | 8 | 16
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Multiple logistic regression modeling used to compute adjusted odds ratios for 12-month follow-up data; Test type: Superiority; p = .037, Regression, Logistic; Adjusted for group differences at baseline and variables associated with differential study retention; Odds Ratio (OR) = 0.25, 95% CI 2-sided [.07 to .92] — Usual care arm is reference group

2. Primary Outcome: Rapid Repeat Pregnancy
Description: Number and percent with any repeat pregnancy by each follow-up time point.
Time Frame: 24 months follow-up
Population: Participants with pregnancy data available at 24 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 55 | 52
Participants | 17 | 24
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .029, Regression, Logistic; Adjusted for any variables that differed between groups at baseline, and variables associated with likelihood of study retention at follow-up; Odds Ratio (OR) = .24, 95% CI 2-sided [.07 to .86] — Usual care arm is reference group

3. Primary Outcome: Rapid Repeat Pregnancy
Description: Number and percent with any repeat pregnancy by each follow-up time point.
Time Frame: 36 months follow-up
Population: Participants with pregnancy data available at 36 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 52 | 48
Participants | 22 | 32
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .017, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = .20, 95% CI 2-sided [.06 to .75] — Usual care arm is the reference group

4. Secondary Outcome: Maternal Parenting Self-esteem Total Score
Description: Total score from the widely used Maternal Self-Report Inventory (MSRI) (Shea E & Tronick EZ, 1988). The measure is comprised of 26 items with response items "completely false", "mainly false", "uncertain or neither true or false", "mainly true", and "completely true." The item response scale ranged from 1-5, with higher scores indicating higher maternal self-esteem. The total score is a sum of all items, thus the minimum/maximum possible scores are 26-130. Higher scores indicate higher maternal self-esteem.
Time Frame: 12-month follow-up
Population: Number that completed the MSRI at 12 months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Young Parents Program Plus Parenting/Life Skills Modules: Modules: These modules were developed using the Ansell-Casey Life Skills Assessment Curriculum and The Women's Negotiation Project Curriculum for Teen Mothers. The Nurturing Curriculum has been shown in our past program to be associated with increased parenting skills, maternal self-esteem and decreased life hassles. The nationally recognized Nurturing Curriculum is integrated with the Ansell-Casey life skills Curriculum and The Women's Negotiation Project Curriculum to help teen mothers develop the skills and communication needs of daily living. The series of five, one-hour long, structured, one-on-one interactive modules aims to help teens build positive, empathetic relationships with their children, while enhancing self-efficacy and increasing the sense of self- worth for parents and children. Domains addressed include child development/discipline, safety, house/money management, social relationships, career planning, substance abuse and community and interpersonal violence.
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 49 | 60
score on a scale | 116.2 (1.8) | 112.8 (1.7)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .217, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 4.75, Standard Error of Mean 3.84

5. Secondary Outcome: Maternal Parenting Self-esteem Total Score
Description: as for outcome 4
Time Frame: 24-month follow-up
Population: Number that completed the MSRI at 24 months follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 57
score on a scale | 112.8 (1.9) | 110.4 (2.4)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .444, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 2.89, Standard Error of Mean 3.77

6. Secondary Outcome: Maternal Parenting Self-esteem Total Score
Description: as for outcome 4
Time Frame: 36-month follow-up
Population: Number that completed the MSRI at 36 months follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 51
score on a scale | 108.5 (2.6) | 99.4 (3.1)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .011, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 9.76, Standard Error of Mean 3.82

7. Secondary Outcome: Parenting Profile - Parent-Child Role Responsibilities
Description: Subscale sten score from the 40-item Adult-Adolescent Parenting Inventory-2 (Bavolek SJ & Keene RG). Min/max score range = 1-10. Higher scores indicate better parenting and lower risk for child maltreatment.
Time Frame: 12-month follow-up
Population: Number that completed the AAPI-2 at 12-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 49 | 60
score on a scale | 5.9 (0.4) | 5.6 (0.3)

8. Secondary Outcome: Parenting Profile - Parent-Child Role Responsibilities
Description: as for outcome 7
Time Frame: 24-month follow-up
Population: Number that completed the AAPI-2 at 24-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 55 | 52
score on a scale | 5.4 (0.4) | 4.8 (0.4)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .758, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = .64, Standard Error of Mean .59

9. Secondary Outcome: Parenting Profile - Parent-Child Role Responsibilities
Description: as for outcome 7
Time Frame: 36-month follow-up
Population: Number that completed the AAPI-2 at 36-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 51
score on a scale | 5.1 (0.3) | 3.7 (0.4)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .024, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 1.36, Standard Error of Mean .60

10. Secondary Outcome: Life Skills Score
Description: Total raw score on Ansell-Casey Life Skills (ACLS) Assessment assessing skills of daily living, communication, and relationships. Min/max score range = 37-111. Higher scores indicate higher life skills.
Time Frame: 12-month follow-up
Population: Number that completed the ACLS at 12-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 49 | 60
score on a scale | 83.0 (2.0) | 81.4 (2.5)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .354, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 2.67, Standard Error of Mean 2.88

11. Secondary Outcome: Life Skills Score
Description: as for outcome 10
Time Frame: 24-month follow-up
Population: Number that completed the ACLS at 24-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 57
score on a scale | 87.0 (2.2) | 83.4 (2.3)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .121, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 4.43, Standard Error of Mean 2.85

12. Secondary Outcome: Life Skills Score
Description: as for outcome 10
Time Frame: 36-month follow-up
Population: Number that completed the ACLS at 36-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 51
score on a scale | 90.6 (2.1) | 87.5 (2.7)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .205, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 3.67, Standard Error of Mean 2.89

13. Secondary Outcome: Depressive Symptoms Score
Description: Total score on the 20-item Centers for Epidemiologic Studies Depression Scale for Children (CES-DC). Min/max score range = 0-60. Higher scores indicate higher depressive symptoms. Scores over 15 indicate significant level of depressive symptoms.
Time Frame: 12-month follow-up
Population: Number that completed the CES-DC at 12-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 49 | 60
score on a scale | 21.2 (1.9) | 17.6 (1.7)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .803, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 0.65, Standard Error of Mean 2.60

14. Secondary Outcome: Depressive Symptoms Score
Description: as for outcome 13
Time Frame: 24-month follow-up
Population: Number that completed the CES-DC at 24-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 57
score on a scale | 18.0 (1.6) | 14.5 (1.2)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .347, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = 2.41, Standard Error of Mean 2.56

15. Secondary Outcome: Depressive Symptoms Score
Description: as for outcome 13
Time Frame: 36-month follow-up
Population: Number that completed the CES-DC at 36-months follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Young Parents Program Plus Parenting/Life Skills Modules | Young Parents Program Usual Care
Number analyzed (Participants) | 58 | 51
score on a scale | 16.4 (1.4) | 17.0 (1.7)
Statistical Analysis 1: Comparison: Young Parents Program Plus Parenting/Life Skills Modules vs Young Parents Program Usual Care; Test type: Superiority; p = .591, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Group by time interaction term coefficie = -1.39, Standard Error of Mean 2.59

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Non Randomized: These are those mothers in the group who choose not to be randomized into the study, or the fathers who participate who are not randomized into the study.
  No intervention: Those in the control group receive the YPP standard of care including comprehensive multi-disciplinary team medical and mental health support and toddler educational family forums during year 2.
- Modules: These modules were developed using the Ansell-Casey Life Skills Assessment Curriculum and The Women's Negotiation Project Curriculum for Teen Mothers. The Nurturing Curriculum has been shown in our past program to be associated with increased parenting skills, maternal self-esteem and decreased life hassles. The nationally recognized Nurturing Curriculum is integrated with the Ansell-Casey life skills Curriculum and The Women's Negotiation Project Curriculum to help teen mothers develop the skills and communication needs of daily living. The series of five, one-hour long, structured, one-on-one interactive modules aims to help teens build positive, empathetic relationships with their children, while enhancing self-efficacy and increasing the sense of self- worth for parents and children. Domains addressed include child development/discipline, safety, house/money management, social relationships, career planning, substance abuse and community and interpersonal violence.
- Control: Patients receive regular standard of care without modules.
  No intervention
Arm/Group | Non Randomized | Modules | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/72 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/72 | 0/68
Other Adverse Events (participants affected / at risk) | 0/12 | 0/72 | 0/68

LIMITATIONS AND CAVEATS:
* Outcomes data were based on self-report, but repeat pregnancies were verified by chart review
* Engaging and retaining teen mothers in the intervention was challenging, but adherence was similar to other teen parenting programs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No